CLINICAL TRIAL: NCT06243263
Title: Postoperative Pain After Bupivacaine Supplementation in Mandibular Fracture Surgery: a Double Blind Controlled Clinical Trial
Brief Title: Postoperative Pain After Bupivacaine Supplementation in Mandibular Fracture Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Yasmine Sanaa, Yasmine Moufida Sanaa , MD, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: T00000228
Record Dates: First submitted 2024-01-27; First posted 2024-02-06 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain; Mandible Fracture; Analgesia; Anesthesia, Local
Keywords: Mandibular Fracture, Postoperative pain, Inferior alveolar nerve block, Analgesia
MeSH Terms: conditions — Pain, Postoperative; Mandibular Fractures; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants with bifocal mandibular fractures will be enrolled in the study (a fracture should be located on the dentate portion of the right hemi-mandible, and a second fracture located on the dentate portion of the left hemi-mandible). Each patient will receive either a right or left inferior alveolar nerve block with bupivacaine.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group BNAI+ (Experimental): Randomization process will be used to preoperatively assign patient's left or right side to receive inferior alveolar nerve block. At the end of the surgery, each patient will receive an inferior alveolar nerve block with 2ml of bupivacaine 0.5% on one side ;the other side will not be injected. This arm include the group of fracture which will receive an inferior alveolar nerve block with bupivacaine.
  All patient will receive during the postoperative period 1 gram of paracetamol each 8 hours.
  Interventions: Drug: Bupivacain
- Group BNAI- (No Intervention): Randomization process will be used to preoperatively assign patient's left or right side to receive inferior alveolar nerve block. At the end of the surgery, each patient will receive an inferior alveolar nerve block with 2ml of bupivacaine 0.5% on one side ;the other side will not be injected. This arm include the group of fracture which will not receive an inferior alveolar nerve block with bupivacaine ( control group).
  All patient will receive during the postoperative period 1 gram of paracetamol each 8 hours.

INTERVENTIONS:
Drug: Bupivacain — At the end of the surgery, after wound closure, an inferior alveolar nerve block with 2ml bupivacaine 0,5 % will be realized.
  Arms: Group BNAI+

SUMMARY:
Pain following open reduction of mandibular fractures is the most reported complaint during the first 24 post-operative hours. The goal of this clinical trial is to evaluate the impact of inferior alveolar nerve block with bupivacaine 0,5% in patients with mandibular fractures.

The main question it aims to answer are:

* Does the inferior alveolar nerve block with bupivacaine reduce the intensity of pain after mandibular fracture surgery?
* Does the inferior alveolar nerve block with bupivacaine decrease the consumption of analgesics during the first 24 postoperative hours?

Participants with bifocal mandibular fractures will be enrolled in the study (a fracture should be located on the dentate portion of the right hemi-mandible, and a second fracture located on the dentate portion of the left hemi-mandible). Each patient will receive either a right or left inferior alveolar nerve block.

The patient:

* Will be asked to estimate the pain score by the numerical rating scale during the first 24 postoperative hours for each fracture.
* They will be given rescue analgesia in case of intense pain. The number of uses of rescue analgesia will be noted.

Researchers will compare a group of fracture that will receive the inferior alveolar nerve block with bupivacaine with a group of fracture that will not receive the inferior alveolar nerve block, to see if regional anesthesia improve postoperative pain management of mandibular fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bifocal mandibular fractures ( with one fracture on the dentate portion of the right hemi-mandible, and a second fracture located on the dentate portion of the left hemi-mandible )
* Proposed for open reduction and internal fixation of their fractures under general anesthesia;
* Having provided their informed and documented consent on a consent form.

Exclusion Criteria:

* Pathological mandibular fractures;
* History of mandibular fractures;
* Patients with bone involvement in the facial skeleton other than the two fractures of the mandibular dentate portion;
* Patients suffering from trigeminal neuralgia;
* Dental care performed in the month preceding the trauma;
* Patients who have not undergone surgical treatment with open reduction and internal fixation of their mandibular fractures;
* Patients on anticoagulants;
* Porphyrias;
* History of malignant hyperthermia;
* Known allergy to local anesthetics;
* Pregnancy or breastfeeding;
* Severe heart failure;
* Atrioventricular conduction disorders;
* Uncontrolled epilepsy;
* Hemostatic disorders;
* Non-cooperative patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-06 (Estimated); Primary Completion 2024-03-04 (Estimated); Study Completion 2024-03-04 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 8 hours post-operatively
  questionnaire with a numerical scale (0 - 10)

SECONDARY OUTCOMES:
Post-operative pain | 2, 4 , 12, 24 hours post-operatively
  questionnaire with a numerical scale (0 - 10)
Adverse effects | 24 hours post-operatively
  questionnaire including the presence or absence of any abnormal sensations, change in taste, nausea, constipation, fever, diaphoresis, vomiting, light-headedness, palpitations, or headache. The notice of an hematoma or in infection at the site of the injection
The number of instances of rescue analgesia | 24 hours post-operatively
  We will record the number of instances of rescue analgesia following the description of intense pain for each hemi-mandible group.

CONTACTS AND LOCATIONS:
Locations (2):
- Tunisia (2):
  - Charles Nicole Hospital, Tunis
  - Charles Nicolle Hospital of Tunis, Tunis